CLINICAL TRIAL: NCT05437107
Title: Mechanism and Intervention Research of Atherosclerosis
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-I2M-1-009
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Atherosclerosis
Keywords: mechanism; biomarker; atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with atherosclerosis are at high risk of future cardiovascular disease. Approximately 70% cardiac death and 50% myocardial infarction (MI) occurred among patients with established coronary artery disease (CAD). These patients have a four to seven-fold risk of fatal or non-fatal MI compared with those without CAD. Current secondary prevention therapy, including statins and anti-platelet therapy have decreased mortality among CHD patients. However, one out of five patients with MI experienced cardiovascular events within one-year of discharge.

This study aims at identifying new risk factors of atherosclerosis, improving risk-stratification among patients with CAD by using novel biomarkers and finally improving outcome and life quality of patients. The investigators will recruit 30000 patients undergoing elective elective coronary angiography and collect baseline characteristics, physical examination, lab test results, angiographic characteristics, etc. Blood sample will also be collected at baseline. Subsequently, two-year follow-up will be done to collect data regarding patients' outcome, including cardiac death, MI, revascularization, medication, etc. Investigators will compare baseline, imaging, blood test results between patients with and without cardiovascular events and identify novel predictors of the occurrence and progression of CAD.

DETAILED DESCRIPTION:
1. Organization of the project This project involves the cooperation between different teams. Principle investigator is responsible for all aspects of the project, including design, executive, monitoring and report of the project. Scientific committee is responsible for the scientific design of the registry, as well as rational design of subsequent studies based on the registry. Data management team will monitor the logic, validity, consistency, completeness of data and provide timely feedback to researchers. Clinical support team and Statistics team are responsible for the medical, and data analysis aspect of the registry respectively.
2. Data quality assurance Data are collected, submitted and stored online to the Informatics Center of Fuwai Hospital. Data are stored and protected managed according to national information security protection law. The following measures are adopted for data quality control. (1) Research staff will only be given access to a password-protected data-entry system after formal training. (2) A real-time, automated algorithm is used to check the logic, range, validity, consistency, completeness of data entered in the system. (3) Approximately 10% of online records are selected randomly and checked against the source documentation. (4) Data management team will check data quality regularly, and ask research staff to review and revise the missing, invalid and illogical data.
3. Data dictionary Data are collected by trained experienced cardiologists and by using standardized definition in accordance with ACC/AHA Task Force on clinical Data Standards and NCDR-CathPCI registry Data Coder's Dictionary, including patient demographics, clinical presentation, medical history, risk factors, physical examination, laboratory results, clinical events, angiographic characteristics and procedural characteristics.
4. Sample size, missing data We didn't set upper limits for sample size and plan to enroll all eligible participants admitted to Fuwai hospital, because we aim to obtain a comprehensive understanding of the management and outcome of patients with suspected CAD and receiving coronary angiography. According to Fuwai Hospital data, number of PCI procedure reached 17798. Therefore we plan to enroll 30000 patients from January 2017 to December 2018.

Several measures will be adopted to manage missing data: (1) "Required" fields are used for key variables during data entry. (2) We conducted pilot testing to identify variables with high rate of missing data, explore possible reasons and improve data collection. (3) Data management team will monitor data quality periodically and send queries to researchers to enter the missing data and check invalid data. (4) During statistical analysis phase, based on the type, pattern and amount of missing data, appropriated methods will be used to handle missing data.

ELIGIBILITY:
Inclusion Criteria:

* Undergo elective coronary angiography in department of cardiology in period of study
* Written informed consent

Exclusion Criteria:

* Age ≤18 years of age
* Unable to sign consent
* Other severe comorbidities with life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suspected of CAD and underwent elective coronary angiogram. Patients have signed written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 2 years
  death, nonfatal myocardial infarction, repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, MD, PhD, Principal Investigator — National Center for Cardiovascular Diseases; Fuwai Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Yuejin Yang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No